CLINICAL TRIAL: NCT01175278
Title: A Pilot Study of Vertebral Augmentation With Kyphoplasty Versus Nonsurgical Management in Multiple Myeloma Patients With Mildly Symptomatic Vertebral Body Compression Fractures
Brief Title: Vertebral Augmentation With Kyphoplasty vs Nonsurgical Mgmt for Vertebral Body Compression Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Medtronics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15839; Pro00000214 (Other: USF Institutional Review Board)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Myeloma
Keywords: vertebral; compression; fracture; VCF; kyphoplasty; spine
MeSH Terms: conditions — Multiple Myeloma; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observation Arm (No Intervention): Patients who are asymptomatic (no symptoms) will participate in the observational portion of the study.
- Balloon Kypholasty (Experimental)
  Interventions: Procedure: Vertebral Augmentation with Balloon Kyphoplasty
- Control Arm (Active Comparator): Non-surgical Management Treatment Group
  Interventions: Other: Non-surgical Treatment

INTERVENTIONS:
Procedure: Vertebral Augmentation with Balloon Kyphoplasty — Two small metal tubes will be inserted through the skin into the collapsed bone. Inflatable bone tamps (balloon catheters) will be inserted through each of these two tubes into the bone. The balloons will be inflated with a liquid that can be seen on xrays (contrast) to return the bone toward its natural shape and create a cavity. The balloons will then be deflated and removed. The cavity in the bone will be filled with bone cement to stabilize the broken backbone.
  Arms: Balloon Kypholasty
Other: Non-surgical Treatment — Non-surgical treatment means the institution of therapies other than cancer chemotherapy and surgical treatment aimed at alleviation of back pain and restoration of decreased function associated with the patient's VCF(s).
  Arms: Control Arm

SUMMARY:
The purpose of this study is to find out how balloon kyphoplasty (surgical repair of the patient's fracture using balloons and bone cement) compares to non-surgical treatment in reducing vertebral compression fractures while providing pain relief and improved function and quality of life.

DETAILED DESCRIPTION:
This is a prospective single center study designed to compare balloon kyphoplasty to non-surgical management (NSM) in the treatment of mildly painful, acute vertebral body compression fractures in multiple myeloma patients. Because of the pilot nature and the small sample size of the study, patient randomization will NOT be stratified. Patients with mildly symptomatic vertebral compression fractures (VCFs) will undergo a 1:1 randomization either balloon kyphoplasty or non surgical management. Randomization assignments will be generated by computer and investigator notified once the patient enrolled.

The observational arm will be compared to each of the other two arms; control and intervention arm using the same outcome variables and statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma (active or smoldering) with mild back pain (Visual Analog Scale [VAS]) ≤ 4 or no back pain (VAS=0) on a stable analgesic regimen) related to vertebral compression fractures (at least one and up to 8 index fractures from T3 to L5) as seen on magnetic resonancy imaging (MRI), computed axial tomography (CT) scan or plain radiographs.
* No major planned spine surgery for at least 6 months following enrollment.
* No evidence of epidural disease or cord compromise on magnetic resonance imaging.
* Life expectancy greater than 6 months.
* Adequate myeloma systemic control (no evidence of active progressive disease). No planned change in chemotherapy regimen for 1 month prior and for at least 1 month following enrollment. Change in dose(s) permitted.
* Adequate hematologic parameters (platelet count≥50,000/μL, and absolute neutrophil count ≥1,000). Platelet transfusions are permitted to increase platelet counts perioperatively.
* Age greater than 21 years and able to understand and sign the informed consent document.

Exclusion Criteria:

* Patients with significant comorbidities (aside from the index fracture or cancer) which would result in an unacceptable surgical risk or patients with contraindications to general or local anesthesia.
* Patients with other primary tumors including primary bone tumors or solitary plasmacytoma at site of the index VCF.
* VCF morphology deemed unsuitable for balloon kyphoplasty (vertebra planum).
* Additional non-kyphoplasty surgical treatment is required for the index fracture.
* Patients with uncontrolled pain related to the VCF (VAS>4, or increasing opioid requirements), or with epidural disease on magnetic resonance imaging. Spinal cord compression , canal compromise and /or spinal instability requiring decompression.
* Patients with a bleeding disorder which cannot be adequately managed perioperatively.
* Patients with pain unrelated to the VCF according to the investigators.
* Patients with estimated survival less than 6 months.
* Known allergy to bone cement or all contrast media used in the treatment of study participants.
* MRI contraindication (e.g., cerebral aneurysm clips, pacemaker, implanted biostimulators, cochlear implants, penile prosthesis).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time to Vertebral Event | Average of 12 months
  Time to vertebral event (composite end point of pain progression, hospitalization for pain, and rescue vertebral augmentation or surgery or radiation therapy as related to an index fracture)
Time to Pain Progression | Average of 12 months
  Time to pain progression defined as the time to the development of pain severity rated greater than 4 on the visual analog scale (VAS) as related to an index fracture

SECONDARY OUTCOMES:
Rate of Vertebral Events | 12 months
  Rate of vertebral events in patients with asymptomatic vertebral compression fracture at 12 months
Rate of Hospitalization | 12 months
  Rate of hospitalization for pain control in patients with asymptomatic or mildly symptomatic vertebral compression fracture at 12 months
Complications of Procedure | Average of 12 months
  Complications of vertebral augmentation
Quality of Life Questionnaire Results | Average of 12 months
  Quality of life as assessed by the Functional Assessment of Cancer Treatment - General (FACT-G) questionnaire in all enrolled patients and Roland Morris disability questionnaire for spine disability
Changes in Pulmonary Function | Average of 12 months
  Changes in pulmonary function testing in patients with thoracic spine vertebral compression fracture
Change in Kyphosis | Average of 12 months
  Change in kyphosis as measured by the Cobb method and change in vertebral collapse by the method of Genant
Prognostic Ability of Bone Biomarkers | Average of 12 months
  Prognostic ability of bone biomarkers for the prediction of vertebral events

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vrionis, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute